CLINICAL TRIAL: NCT01577680
Title: An Open-label, Non-randomized, Pharmacokinetic and Safety Study of Single Dose GSK573719 + GW643444 (VI) Combination and Repeat Doses of GSK573719 in Healthy Subjects and in Subjects With Moderate Hepatic Impairment
Brief Title: A Study to Assess the Effects of GSK573719/VI Combination and GSK573719 Monotherapy in Subjects With Moderate Hepatic Impairment and Matched Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 114637
Record Dates: First submitted 2012-03-29; First posted 2012-04-16 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: healthy subjects; pharmacokinetics; vilanterol; tolerability; safety; hepatic impairment; GW642444; GSK573719
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — vilanterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Hepatic Impairment (Experimental): Approximately 9 subjects will complete each of these treatment arms
  Interventions: Drug: Inhaled GSK573719/vilanterol; Drug: Inhaled GSK573719
- Matched Healthy Volunteers (Experimental): Matched to the moderate hepatic impairment subjects based on gender, ethnicity, body mass index (+/-15%) and age (+/-5 years) Approximately 9 subjects will complete each of these treatment arms
  Interventions: Drug: Inhaled GSK573719/vilanterol; Drug: Inhaled GSK573719

INTERVENTIONS:
Drug: Inhaled GSK573719/vilanterol — All subjects will receive a single dose of GSK573719/VI (125mcg/25mcg) in Treatment Period 1
Drug: Inhaled GSK573719 — All subjects will receive GSK573719 (125mcg) once daily for seven days in Treatment Period 2

SUMMARY:
This study will assess the safety and pharmacokinetics of GSK573719 and GSK573719/vilanterol combination in healthy subjects and subjects with moderate hepatic impairment. The results of this study will provide guidance on the use of the product in patients with hepatic impairment.

DETAILED DESCRIPTION:
GSK573719 is being developed as a monotherapy and in combination with vilanterol for the treatment of Chronic Obstructive Pulmonary Disease (COPD). This study will assess the pharmacokinetics and safety of inhaled GSK573719/ vilanterol (VI) and GSK573719 in healthy subjects and in subjects with moderate hepatic impairment. Nine subjects with moderate hepatic impairment will be recruited, together with nine matched healthy volunteers.

There is a possibility that when used by patients with impaired hepatic function the pharmacokinetics of inhaled GSK573719 or GSK572719/VI may be altered. The results of this study will therefore provide guidance on the use of GSK573719 and GSK573719/VI in moderate hepatically impaired patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 70 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea Child-bearing potential and is abstinent or agrees to use one of the contraception methods listed in the protocol

* Body weight of greater than or equal to 45 kg and body mass index within the range 18 - 33 kg/m2 (inclusive).
* Single QTcF less than 450 msec; or QTc less than 480 msec in subjects with Bundle Branch Block.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form Healthy Subjects
* ALT, alkaline phosphatase and bilirubin less than or equal to 1.5x Upper Limit of Normal (ULN)
* Healthy as determined by a responsible and experienced physician Hepatically Impaired Subjects
* Moderately hepatically impaired - subjects must have a known medical history of liver disease with or without a known history of alcohol abuse, and a Child-Pugh score of 7-9 points
* Subjects with no significant abnormality, apart from impaired hepatic function and related symptoms, or clinical examination.

Exclusion Criteria:

* Suffered a lower respiratory tract infection in the 4 weeks before the screening visit.
* A supine mean heart rate outside the range 40-90 beats per minute (BPM) at screening.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females
* Subjects with smoking history of greater than 10 cigarettes per day or regular use of tobacco- or nicotine-containing products, within 6 months prior to screening.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* The subject is unable to use the novel dry powder inhaler correctly Healthy Subjects
* Subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism or excretion of drugs or any previous gastrointestinal (GI) surgery condition which the investigator considers sufficiently significant to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units for males or 14 units for females
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication

Hepatically impaired subjects:

* If in the opinion of the examining physician, an unstable cardiovascular, renal, pulmonary, endocrine, metabolic, neurological, haematological or gastrointestinal condition is present or any other significant medical condition which the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* Severe ascities (Child-Pugh ascites score of 3) upon clinical exam, including physical exam and abdominal ultrasound at screening. Subjects identified to have moderate ascities by ultrasound examination may be included at the discretion of the Investigator with prior agreement from the sponsor.
* History of oesophageal bleeding within the last 6 months before dosing.
* Significant hepatic encephalopathy, degree of CNS impairment or other signs of hepatic function deterioration which the investigator considers sufficiently serious to interfere with the informed consent, conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* Patients at risk of requiring a transfusion during the study period, or has haemoglobin less than 9 g/dL
* Evidence of current significant infection
* Subjects who develop symptoms such as infections or haemorrhage between screening and dosing must not be included in the study
* Fluctuating or rapidly deteriorating hepatic function
* Subjects with significant renal insufficiency as defined by estimated creatinine clearance of less than 50 ml/min, using the Cockcroft and Gault equation
* Subjects with a diagnosis of primary biliary disease such as cholestasis or sclerosing cholangitis
* Subjects who need to take any concomitant medication, either prescribed or overthe- counter, which may in the opinion of the Investigator, interfere in any way with the study procedure or be a safety concern. In particular subjects taking medications that significantly inhibit P450 CYP3A4 (e.g. ketoconazole) must not be included in this study
* Subjects who, within the past six months, have had a history of significant drug abuse or alcohol abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03-05 (Actual); Primary Completion 2012-06-29 (Actual); Study Completion 2012-06-29 (Actual)

PRIMARY OUTCOMES:
GSK573719 and vilanterol pharmacokinetics | Treatment Period 1: Pre-dose, 5 mins, 15 mins, 30 mins, 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 16 hrs, 24 hrs
  Including AUC(0-t), AUC(0-t'), Cmax, tmax, AUC(0-24), AUC(0-infinity), tlast, t1/2 (following single dose administration)
GSK573719 pharmacokinetics | Treatment Period 2 (Day 1 and 7): Pre-dose, 5 mins, 15 mins, 30 mins, 1 hr, 2hrs, 4 hrs, 8 hrs, 12hrs, 16 hrs, 24 hrs (and 36 hrs on Day 7 only)
  Including AUC(0-t), AUC(0-t'), Cmax, tmax, AUC(0-24), AUC(0-infinity), tlast, t1/2 (following single and repeat dose administration)

SECONDARY OUTCOMES:
Urine pharmacokinetics for GSK573719 (Treatment Period 1) | 0-4hrs, 4-8hrs, 8-12hrs and 12-24hrs
  Including amount excreted in urine in 24 hrs (following single dose administration)
Urine pharmacokinetics for GSK573719 (Treatment Period 2) | Days 1 and 7: 0-4hrs, 4-8hrs, 8-12hrs, 12-24hrs (and 24-36hrs on Day 7 only)
  Including amount excreted in urine in 24 hrs (following single and repeat dose administration)
Measurement of vital signs | Screening (up to 21 days before dosing), Treatment Period 1 and Treatment Period 2 (Day 1 and 7): pre-dose, 5 mins, 15 mins, 30 mins, 1 hr, 4 hrs, 12 hrs, 24 hrs, Follow-up (7 to 14 days after last dose)
  Including systolic and diastolic blood pressure and heart rate
Adverse Events | Adverse events will be recorded from the start of dosing to follow-up (7 to 14 days after last dose), an average expected duration of 4 weeks
Clinical Laboratory Safety Tests | Screening (up to 21 days before dosing), Treatment Period 1: pre-dose, 24 hrs, Treatment Period 2 (Day 1 and 7): pre-dose, 24 hrs, Day 4 hepatic subjects only, Follow-up (7 to 14 days after last dose)
  Including haematology, clinical chemistry and urinalysis tests
12-lead ECG measurements | Screening (up to 21 days before dosing), Treatment Period 1 and Treatment Period 2 (Day 1 and 7): pre-dose, 5 mins, 15 mins, 30 mins, 1 hr, 4hrs, 12hrs, 24hrs

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Budapest, Hungary
- GSK Investigational Site, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114637 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114637?search=study&search_terms=114637#rs
- Available data/document: Statistical Analysis Plan: 114637 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114637 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114637 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114637 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114637 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114637 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114637 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register